CLINICAL TRIAL: NCT04267198
Title: Intention Treatment for Anomia: Investigating Dose Frequency Effects and Predictors of Treatment Response to Improve Efficacy and Clinical Translation
Brief Title: Intention Treatment for Anomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N3093-R
Record Dates: First submitted 2020-02-04; First posted 2020-02-12 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Aphasia; Stroke
Keywords: aphasia; language; rehabilitation; speech-language pathology
MeSH Terms: conditions — Aphasia; Stroke; Language

STUDY DESIGN:
Intervention Model Description: Delayed-start controlled trial with stratification across two groups (massed-INT, distributed-INT) based on severity of word retrieval deficits.
Who Masked: Outcomes Assessor
Masking Description: Assessments will be conducted by study staff blind to treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Massed Intention Treatment (massed-INT) (Active Comparator): Participants will receive 30 hours of Intention Treatment (INT) over 3 weeks.
  Interventions: Behavioral: Intention Treatment for Anomia
- Distributed Intention Treatment (distributed-INT) (Active Comparator): Participants will receive 30 hours of Intention Treatment (INT) over 12 weeks.
  Interventions: Behavioral: Intention Treatment for Anomia

INTERVENTIONS:
Behavioral: Intention Treatment for Anomia — Word retrieval treatment for aphasia that engages right hemisphere intention mechanisms using a left-hand circular gesture.

SUMMARY:
Every year approximately 15,000 Veterans are hospitalized for stroke, and up to 40% of those Veterans will experience stroke-related language impairment (i.e., aphasia). Stroke-induced aphasia results in increased healthcare costs and decreased quality of life. As the population of Veterans continues to age, there will be an increasing number for Veterans living with the aphasia and its consequences. Those Veterans deserve to receive aphasia treatment designed to facilitate the best possible outcomes. In the proposed study, the investigators will investigate optimal treatment intensity and predictors of treatment response for a novel word retrieval treatment. The knowledge the investigators gain will have direct implications for the selecting the right treatment approach for the right Veteran.

DETAILED DESCRIPTION:
Difficulty retrieving words is one of the most common language complaints in individuals with stroke-induced aphasia. The negative consequences related to word retrieval impairment include increased health care costs and decreased quality of life. A variety of treatment approaches exist to improve word retrieval, and most of the treatments result in immediate improvement on trained words. However, long-term improvement and improvement on untrained words or behaviors is less common. Additionally, the investigators currently know very little about optimal treatment administration parameters, and the investigators know even less about predictors of treatment response. To make the best use of the limited clinical resources available for aphasia treatment, and to maximize outcomes for Veterans with aphasia, the investigators must: 1) develop clinically translatable treatments that yield widespread and lasting effects and 2) develop clinically accessible ways of identifying who will acquire benefit from a specific treatment approach. This study takes on these two challenges by investigating dose frequency (massed vs. distributed practice) effects and by identifying the language, cognitive and neural predictors of response to Intention treatment (INT), a novel word retrieval treatment. Specifically, the investigators will address the following aims:

Aim 1: To investigate dose frequency effects on maintenance and generalization of INT gains. Outcome measure: Word retrieval accuracy for trained and untrained words.

Aim 2: To identify the language and cognitive variables that predict response to m-INT vs. d-INT. Outcome measure: Language and cognitive ability as measured by standardized assessments.

Aim 3: To identify the neural predictors of response to m-INT vs. d-INT. Outcome measure: Tissue health and task activation location as measured by structural and functional MRI.

ELIGIBILITY:
Inclusion Criteria:

* English as primary language
* > 6 months post-onset a left-hemisphere stroke. Multiple strokes are acceptable as long as they are confined to the left hemisphere.
* Diagnosis of aphasia
* Presence of word retrieval deficits
* Adequate comprehension as judged by ability to complete two-step commands on the Western Aphasia Battery.

Exclusion Criteria:

* Severe apraxia of speech or dysarthria
* Clinically significant depression
* For MRI safety: implanted medical devices, metal in the body and claustrophobia.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Number of correctly named pictures | Through study completion, an average of 6 months; Change from baseline to 3 weeks (post massed-INT) or 12 weeks (post distributed-INT), change at 3 months post-treatment, change at 6 months post-treatment
  Change in the ability to correctly name 10 trained and 10 untrained pictures will be measured at 4 time points
Number of correctly generated category members | Through study study completion, an average of 6 months; Change from baseline to 3 weeks (post m-INT) or 12 weeks (post d-INT), change at 3 months post-treatment, change at 6 months post-treatment
  Change in the ability to correctly name 5 trained and 5 untrained category members will be measured at 4 time points
Western Aphasia Battery | Baseline
  This standardized assessment will be administered at baseline to investigate language predictors of treatment outcome
Boston Naming Test | Baseline
  This standardized assessment will be administered at baseline to investigate language predictors of treatment outcome
Test of Everyday Attention | Baseline
  This standardized assessment will be administered at baseline to investigate cognitive predictors of treatment outcome.
Brief Visuospatial Memory Test-Revised | Baseline
  This standardized assessment will be administered at baseline to investigate cognitive predictors of treatment outcome.
Hopkins Verbal Learning Test-Revised | Baseline
  This standardized assessment will be administered at baseline to investigate cognitive predictors of treatment outcome.
Digit Span Backwards | Baseline
  This standardized assessment will be administered at baseline to investigate cognitive predictors of treatment outcome.
Delis-Kaplan Executive Function System (D-KEFS) Sorting | Baseline
  This standardized assessment will be administered at baseline to investigate cognitive predictors of treatment outcome.
Structural MRI scan | Baseline
  Tissue health (from structural scan) will be obtained at baseline to investigate neural predictors of treatment outcome.
Functional MRI scan | Baseline
  Task-based activation location (from functional MRI scans) will be obtained at baseline to investigate neural predictors of treatment outcome.

SECONDARY OUTCOMES:
Delis-Kaplan Executive Function System (D-KEFS) Trails | Baseline
  This standardized assessment will be administered at baseline to investigate cognitive predictors of treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Rodriguez, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT04267198/ICF_000.pdf